CLINICAL TRIAL: NCT06543537
Title: Pilot Randomized Controlled Trial of a Collaborative Agenda-setting Intervention (CASI) for Patients With Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rachel Pozzar, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-358; K23NR020219 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma
Keywords: Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: CASI Intervention (Experimental): Enrolled patients and caregivers will complete:
  * Audio recorded baseline visit
  * CASI via mobile device, laptop, or desktop computer 1 week prior to CASI visit 1
  * Audio recorded CASI visit 1
  * CASI via mobile device, laptop, or desktop computer 1 week prior to CASI visit 2
  * Audio recorded CASI visit 2
  * CASI via mobile device, laptop, or desktop computer 1 week prior to CASI visit 3
  * Audio recorded CASI visit 3
  * End of study visit
  For each enrolled patient, enrolled clinicians will complete:
  * Audio recorded baseline visit
  * Audio recorded CASI visit 1
  * Audio recorded CASI visit 2
  * Audio recorded CASI visit 3
  Enrolled clinicians will also complete:
  * Baseline visit, one time
  * End of study visit, one time
  Interventions: Behavioral: Collaborative Agenda-Setting Intervention
- Arm 2: Control (No Intervention): Enrolled patients and caregivers will complete:
  * Audio recorded baseline visit
  * Audio recorded visit 1 will proceed according to usual, oncology care
  * Audio recorded visit 2 will proceed according to usual, oncology care
  * Audio recorded visit 3 will proceed according to usual, oncology care
  * End of study visit
  For each enrolled patient, enrolled clinicians will complete:
  * Audio recorded baseline visit
  * Audio recorded visit 1 will proceed according to usual, oncology care
  * Audio recorded visit 2 will proceed according to usual, oncology care
  * Audio recorded visit 3 will proceed according to usual, oncology care
  Enrolled clinicians will also complete:
  * Baseline visit, one time
  * End of study visit, one time

INTERVENTIONS:
Behavioral: Collaborative Agenda-Setting Intervention — A collaborative agenda-setting intervention (CASI) to promote patient-centered communication, set agendas for discussion at in-clinic visits, increase discussion of psychosocial concerns, and reduce clinician burden. The intervention is integrated into the patient portal and electronic health record. Prior to a clinic visit, the intervention elicits patients' and caregivers' preferences and concerns, then communicates this information to clinicians. Patients, caregivers, and clinicians receive communication resources, while patients and caregivers receive tailored educational materials and navigation to supportive care services.
  Other Names: CASI
  Arms: Arm 1: CASI Intervention

SUMMARY:
This research is being done to test a new communication tool for people with ovarian cancer, caregivers, and clinicians.

The name of the intervention in this research study is:

-Collaborative Agenda-Setting Intervention (CASI)

DETAILED DESCRIPTION:
This two-arm, parallel group-randomized research study is to test a new communication tool (CASI) for people with ovarian cancer, caregivers, and clinicians. This is a pilot feasibility study, which means this is the first time researchers are studying CASI. Clinicians will be randomized into one of the two study groups, Arm 1 or Arm 2, and patients and caregivers will be enrolled in the study arm to which their clinician has been randomized.

The research study procedures include screening for eligibility, audio recorded clinic visits, and questionnaires.

Participation in this research study is expected to last for up to 12 weeks for patients and caregivers, and for up to 52 weeks for clinicians.

It is expected that up to 112 people will take part in this research study, including up to 50 patients, 50 caregivers, and 12 clinicians (six dyads).

The National Institute for Nursing Research is supporting this research by providing funding.

ELIGIBILITY:
Participant Inclusion Criteria:

* At least 18 years old
* Able to speak, understand, and respond to questions written in English
* Willing to be audio recorded
* Have a diagnosis of advanced ovarian cancer (defined as stage III, stage IV, or recurrent disease)
* Be under the care of a participating clinician dyad
* Be scheduled for chemotherapy during the recruitment period
* Be signed up or willing to sign up for Patient Gateway

Caregiver Inclusion Criteria:

* At least 18 years old
* Able to speak, understand, and respond to questions written in English
* Willing to be audio recorded
* Be a family member, partner, or friend of a patient participant with whom the patient participant discusses their cancer care

Clinician Inclusion Criteria:

* Be employed at DFCI as an oncologist, nurse practitioner, or physician assistant
* Take care of at least 4 patients per month with advanced ovarian cancer (defined as stage III, stage IV, or recurrent disease) in the outpatient setting

Participant Exclusion Criteria:

* Age of <18 years
* Unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate | Pre-consent
  The proportion of approached participants that are enrolled. Feasibility of an efficacy trial is defined as ≥60% enrollment among approached participants.

SECONDARY OUTCOMES:
Acceptability of Intervention | Approximately 12 (patient and caregiver participants) and 52 (clinician participants) weeks after enrollment
  Feasibility of an efficacy trial is defined as a mean Acceptability of Intervention Measure score of ≥4.0 among participants in the intervention group. The Acceptability of Intervention Measure is a four-item questionnaire rated on a 5 point Likert-type scale from 5 "Strongly Agree" to "1 Strongly Disagree" with a total scores range of 4 to 20. A higher score represents greater intervention acceptability.
Proportion of Participant-Rated Intervention Helpfulness | Approximately 12 (patient and caregiver participants) and 52 (clinician participants) weeks after enrollment
  Feasibility of an efficacy trial is defined as ≥60% of participants in the intervention group agreeing with the survey item "the CASI was helpful to me."
Proportion of Participant-Rated Intervention Burden | Approximately 12 (patient and caregiver participants) and 52 (clinician participants) weeks after enrollment
  Feasibility of an efficacy trial is defined as ≤20% of participants in the intervention group agreeing with the survey item "the CASI placed a considerable burden on me."
Change in the Functional Assessment of Cancer Therapy - General (FACT-G) Score from Baseline to 12 Weeks (Arm 1) | Baseline and 12 weeks after enrollment
  Defined as the numeric proportion of participants that experience a clinically meaningful improvement in health-related quality of life from baseline to follow-up. A clinically meaningful improvement is defined as an increase of ≥4 points in the Functional Assessment of Cancer Therapy - General (FACT-G) total score. The FACT-G is a 27-item questionnaire rated on a 5 point Likert-type scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 108. A higher score represents greater participant well-being.
Change in FACT-G Score from Baseline to 12 Weeks (Arm 2) | Baseline and 12 weeks after enrollment
  Defined as the numeric proportion of patient participants that experience a clinically meaningful improvement in health-related quality of life from baseline to follow-up. A clinically meaningful improvement is defined as an increase of ≥4 points in the FACT-G total score.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pozzar, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu